CLINICAL TRIAL: NCT05028023
Title: Effects of Apneic Oxygenation in Regional Cerebral Oxygen Saturation rSO2 During Tracheal Dilatation Procedures in Pediatric Patients (With Acquired Tracheal Stenosis). Innovation and Safety of the Technique
Brief Title: Tracheal Dilatation in Pediatric Patients With Acquired Tracheal Stenosis, and the Effects of Apneic Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, IORDANIDOU DESPOINA, MD, Pediatric Anesthetist, Senior Consultant, Anesthesiology Dpt, Hippokratic General Hospital Thessaloniki, Greece, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4637/25-06-2019
Record Dates: First submitted 2021-08-05; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Apnea+Hypopnea; Tracheal Dilatation; Igel; Tracheal Stenosis; Cerebral Hypoxia; Pediatric Respiratory Diseases
Keywords: Apneic oxygenation; Tracheal stenosis; Tracheal dilatation by Balloon Catheter; i-Gel; Regional cerebral oxygen saturation rSO2 by NIRS; Peripheral oxygen saturation SpO2; Partial pressure of arterial oxygen PaO2; Partial pressure of arterial carbon dioxide PaCO2
MeSH Terms: conditions — Ige Responsiveness, Atopic; Tracheal Stenosis; Hypoxia, Brain

STUDY DESIGN:
Intervention Model Description: This single arm Interventional Study is a comparative clinical trial with the form of before and after intervention (apneic oxygenation), in every participant. During the phases of before and after intervention, parameters of regional cerebral oxygen saturation, peripheral oxygen saturation, arterial blood gases and haemodynamics are recorded in both conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with tracheal stenosis undergoing tracheal balloon dilatation (Experimental): Pediatric patients with severe to median acquired tracheal stenosis undergoing tracheal balloon dilatation, and the effects of apneic oxygenation on regional cerebral oxygen saturation rSO2, pulse oximetry SpO2, and arterial oxygen partial pressure PaO2
  Interventions: Biological: Apneic oxygenation - supplemental high flow oxygen administration by an apneic way

INTERVENTIONS:
Biological: Apneic oxygenation - supplemental high flow oxygen administration by an apneic way — In pediatric patients undergoing tracheal balloon dilatation, oxygenation maintenance is essential, while induction in anesthesia, cessation of spontaneous ventilation by neuromuscular relaxant and pediatric i-gel placement are necessary for access to trachea. After i-Gel placement controlled ventilation with 100% oxygen is initiated. Pediatric bronchoscope and balloon dilatation catheter are advanced into trachea to the stenotic area. Overall dilatation duration is 2,5-3minutes, while the balloon is inflated for 60sec. Every dilatation cession consists of three dilatations. First dilatation is performed without oxygen enrichment. During second and third dilatation, a nelaton catheter, connected with high oxygen flow, is advanced into i-Gel canal, together with bronchoscope and balloon catheter. Effects of no oxygenation and apneic oxygenation in regional cerebral oxygen saturation rSO2, pulse oximetry SpO2, arterial blood gases and haemodynamics are recorded and compared.

SUMMARY:
The study presents an alternative method of tracheal dilatation in pediatric patients with acquired tracheal stenosis. Dilatation is performed by the use of balloon catheter connected with manometer, that is bronchoscopic guided into trachea in the stenotic area, through the wide canal of supraglottic device i-Gel. Every dilatation cession consists of three consequent tracheal balloon dilatations of maximum 3 minutes duration each, followed by 10-15minutes interval of controlled ventilation. The balloon is inflated for 60 seconds to reach predefined pressure, and then deflated. This method is minimal traumatic for tracheal mucosa, and application of several dilatation procedures every 2-3months, in pediatric patients with acquired tracheal stenosis, may lead to a relative reopening of trachea and recession of clinical symptoms.For the right performance of the dilatation procedure, patients receive general anesthesia with cessation of spontaneous ventilation. During procedure, controlled ventilation-oxygenation is impossible, because the i-Gel canal is occupied by bronchoscope and balloon catheter, so patients will remain apneic for a short period of time. For pediatric patients is important to perform proper preoxygenation prior to procedure, and to maintain oxygenation as long as possible during procedure. This is achieved by application of apneic oxygenation, through a small catheter, connected to high flow oxygen. Participants are exposed during first dilation to no oxygenation, while during second and third dilatation to apneic oxygenation. Aim of the study is to investigate primarily whether application of apneic oxygenation, in pediatric patients during tracheal balloon dilatation, maintains regional cerebral oxygen saturation rSO2 in significant higher levels, compared with no application of oxygenation. rSO2 levels are a sensitive index of oxygenation efficacy of the brain, accordingly this refers to a safe procedure. Secondary issues are whether application of apneic oxygenation maintains pulse oximetry SpO2 and artierial oxygen partial pressure PaO2 in higher levels, and what are the effects on arterial carbon dioxide partial pressure PaCO2 and on haemodynamic parameters (heart rate, blood pressure), compared with no application of apneic oxygenation.

DETAILED DESCRIPTION:
The study is taking place in the Bronchoscopy Unit of the 3rd Pediatric Dpt of the Aristotles University of Thessaloniki, in the area of the Operating Rooms in the Hippokratic General Hospital of Thessaloniki, Greece. The procedure of tracheal balloon dilatation was developed and performed in Hippokratic General Hospital of Thessaloniki, Greece, for the last three years. From October 2020, pediatric patients are recruited and enrolled in this study, according to specific criteria, set by the Collaborators of the Pulmonology and Bronchoscopy Unit of the 3rd Pediatric Dpt of Aristotles University of Thessaloniki, Greece. Prior to the dilatation procedure, following steps are necessary, performed by the Principal Investigator:

1.detailed preanesthetic evaluation of the participant, for recognition of clinical signs or pathology, that can complicate the procedure and jeopardize health status 2. written informed consents from parents/caregivers, for anesthesia procedure, for tracheal dilatation procedure, and for participation in the study. All recordings during procedures are performed by the Principal Investigator, and double checked by two Collaborators.In cases of appearance of adverse events during the procedure (i.e. severe desaturation, anaphylactic reaction, severe bronchospasm), it is automatically discontinued, advanced life support is initiated, anesthesia is terminated, and participants are closely monitored during recovery.

Sample size calculation was performed according to G* power analysis 3.1.9.2. and the Means test: for extraction of results is necessary to record at least five different pediatric patients, who will undergo at least four tracheal dilatation cessions.

For statistical analysis, quantitative variables will be described as median values and standard deviation (or IQR), qualitative variables as frequencies and percentages, while significancy level will be defined as <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Persistent clinical signs of inspiratory stridor, combined with high pitched cry, hoarse voice, persistent cough or recurrent inspiratory tract infections
* Bronchoscopic conferment of tracheal stenosis from the subglottic area to the area above carina
* Maintenance of clinical symptoms despite intensive and long drug therapy with inhalational steroids, adrenalin or salbutamol
* Urgent need for expansion of trachea, because of risk of full obstruction of trachea

Exclusion Criteria:

* children with haemodynamic instability prior or during the procedure
* children with active respiratory tract infection
* children with low hemoglobin levels - anemia
* children with physical status, according to the American Society of Anesthesiologists, III and IV
* parents who refuse the participation of their children in the study and to sign the informed consent

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in regional cerebral oxygen saturation rSO2 between first and second tracheal balloon dilatation procedure in children | Changes in regional cerebral oxygen saturation rSO2 between end and strart of first/second tracheal dilatation procedure
  Evaluation of changes in regional cerebral oxygen saturation rSO2, measured by Near InfraRed Spectroscopy NIRS, between end and start of 1st tracheal dilatation procedure in children, where no apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in rSO2, between 1st and 2nd procedure. A greater change (decrease) in regional cerebral oxygen saturation rSO2, in the case of no apneic enrichment, compared to apneic oxygenation application, is expected.
Comparison of changes in regional cerebral oxygen saturation rSO2 between first and third tracheal balloon dilatation procedure in children | Changes in regional cerebral oxygen saturation rSO2 between end and strart of first/third tracheal dilatation procedure
  Evaluation of changes in regional cerebral oxygen saturation rSO2, measured by Near InfraRed Spectroscopy NIRS, between end and start of 1st tracheal dilatation procedure in children, where no apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in rSO2, between 1st and 3rd procedure. A greater change (decrease) in regional cerebral oxygen saturation rSO2, in the case of no apneic enrichment, compared to apneic oxygenation application, is expected.
Comparison of changes in regional cerebral oxygen saturation rSO2 between second and third tracheal balloon dilatation procedure in children | Changes in regional cerebral oxygen saturation rSO2 between end and strart of second/third tracheal dilatation procedure
  Evaluation of changes in regional cerebral oxygen saturation rSO2, measured by Near InfraRed Spectroscopy NIRS, between end and start of 2nd and 3rd tracheal dilatation procedure in children, where in both cases apneic oxygenation is applied, and comparison of changes in rSO2, between 2nd and 3rd procedure. No change in regional cerebral oxygen saturation rSO2, between 2nd and 3rd procedure is expected.

SECONDARY OUTCOMES:
Comparison of changes in pulse oximetry - oxygen saturation SpO2 between first and second tracheal dilatation procedure in children | Changes in pulse oximetry SpO2 between end and start of first/second tracheal dilatation procedure in children
  Evaluation of changes in pulse oximetry - oxygen saturation SpO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in SpO2 between 1st and 2nd tracheal balloon dilatation in children. Higher oxygen saturation SpO2 levels, in the case of apneic oxygenation application, compared to no oxygen enrichment, are expected.
Comparison of changes in pulse oximetry - oxygen saturation SpO2 between first and third tracheal dilatation procedure in children | Changes in pulse oximetry SpO2 between end and start of first/third tracheal dilatation procedure in children
  Evaluation of changes in pulse oximetry - oxygen saturationSpO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in SpO2 between 1st and 3rd tracheal balloon dilatation in children. Higher oxygen saturation SpO2 levels, in the case of apneic oxygenation application, compared to no oxygen enrichment, are expected.
Comparison of changes in arterial oxygen partial pressure PaO2 between first and second tracheal dilatation procedure in children | Changes of arterial oxygen partial pressure PaO2 between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in arterial oxygen partial pressure PaO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PaO2 between 1st and 2nd tracheal balloon dilatation in children. Higher arterial oxygen partial pressure PaO2 levels, in the case of apneic oxygenation application, compared to no oxygen enrichment, are expected.
Comparison of changes in arterial oxygen partial pressure PaO2 between first and third tracheal dilatation procedure in children | Changes of arterial oxygen partial pressure PaO2 between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in arterial oxygen partial pressure PaO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PaO2 between 1st and 3rd tracheal balloon dilatation in children. Higher arterial oxygen partial pressure PaO2 levels, in the case of apneic oxygenation application, compared to no oxygen enrichment, are expected.
Comparison of changes in arterial carbon dioxide partial pressure PaCO2 between first and second tracheal dilatation procedure in children | Changes of arterial carbon dioxide partial pressure PaCO2 between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in arterial carbon dioxide partial pressure PaCO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PaCO2 between 1st and 2nd tracheal balloon dilatation in children. High arterial carbon dioxide partial pressure PaCO2 levels, in both no apneic and apneic oxygenation application cases are expected, and the rate of PaCO2 increase depends on the duration of apnea.
Comparison of changes in arterial carbon dioxide partial pressure PaCO2 between first and third tracheal dilatation procedure in children | Changes of arterial carbon dioxide partial pressure PaCO2 between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in arterial carbon dioxide partial pressure PaCO2 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PaCO2 between 1st and 3rd tracheal balloon dilatation in children. High PaCO2 levels, in both no apneic and apneic oxygenation application cases are expected, and the rate of arterial carbon dioxide partial pressure PaCO2 increase depends on the duration of apnea.
Comparison of changes in acid-base balance PH between first and second tracheal dilatation procedure in children | Changes in acid-base balanc PH between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in acid-base balanc PH between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PH between 1st and 2nd tracheal balloon dilatation in children. An equal decrease in acid-base balanc PH, in both no apneic and apneic oxygenation application cases is expected, and the rate of this decrease depends on the duration of apnea and the subsequent arterial carbon dioxide partial pressure PaCO2 increase.
Comparison of changes in acid-base balance PH between first and third tracheal dilatation procedure in children | Changes in acid-base balance PH between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in acid-base balance PH between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in PH between 1st and 3rd tracheal balloon dilatation in children. An equal decrease in acid-base balance PH, in both no apneic and apneic oxygenation application cases is expected, and the rate of this decrease depends on the duration of apnea and the subsequent arterial carbon dioxide partial pressure PaCO2 increase.
Comparison of changes in Bicarbonate plasma levels HCO3, between first and second tracheal dilatation procedure in children | Changes in Bicarbonate plasma levels HCO3 between end and start of first/second tracheal balloon dilatation procedure in childre
  Evaluation of changes in Bicarbonate plasma levels HCO3 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in HCO3 levels between 1st and 2nd tracheal balloon dilatation in children. An equal minor decrease in Bicarbonate plasma levels HCO3, in both no apneic and apneic oxygenation application cases is expected, and the rate of this decrease depends on the duration of apnea and the subsequent acid-base balance PH decrease.
Comparison of changes in Bicarbonate plasma levels HCO3, between first and third tracheal dilatation procedure in children | Changes in HCO3 between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in Bicarbonate plasma levels HCO3 between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in HCO3 levels between 1st and 3rd tracheal balloon dilatation in children. An equal minor decrease in Bicarbonate plasma levels HCO3, in both no apneic and apneic oxygenation application cases is expected, and the rate of this decrease depends on the duration of apnea and the subsequent acid-base balance PH decrease.
Comparison of changes in Lactate plasma levels Lac, between first and second tracheal dilatation procedure in children | Changes in Lactate plasma levels Lac between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in Lactate plasma levels Lac between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Lac plasma levels between 1st and 2nd tracheal balloon dilatation in children. No changes in Lactate plasma levels Lac, in both no apneic and apneic oxygenation application cases are expected.
Comparison of changes in Lactate plsama levels Lac, between first and third tracheal dilatation procedure in children | Changes in Lactate plasma levels Lac between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in Lactate plasma levels Lac between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Lac plasma levels between 1st and 3rd tracheal balloon dilatation in children. No changes in Lactate plasma levels Lac, in both no apneic and apneic oxygenation application cases are expected.
Comparison of changes in Heart Rate, between first and second tracheal dilatation procedure in children | Changes in Heart Rate between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in Heart Rate between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Heart Rate between 1st and 2nd tracheal balloon dilatation in children. No significant changes in Heart Rate, in both no apneic and apneic oxygenation application cases are expected, although lack of oxygen in children leads to bradycardia.
Comparison of changes in Heart Rate, between first and third tracheal dilatation procedure in children | Changes in Heart Rate between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in Heart Rate between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Heart Rate between 1st and 3rd tracheal balloon dilatation in children. No significant changes in Heart Rate, in both no apneic and apneic oxygenation application cases are expected, although lack of oxygen in children leads to bradycardia.
Comparison of changes in Systolic Blood Pressure, between first and second tracheal dilatation procedure in children | Changes in Systolic Blood Pressure between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in Systolic Blood Pressure between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Systolic Blood Pressure between 1st and 2nd tracheal balloon dilatation in children. No significant changes in Systolic Blood Pressure, in both no apneic and apneic oxygenation application cases are expected.
Comparison of changes in Systolic Blood Pressure, between first and third tracheal dilatation procedure in children | Changes in Systolic Blood Pressure between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in Systolic Blood Pressure between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Systolic Blood Pressure between 1st and 3rd tracheal balloon dilatation in children. No significant changes in Systolic Blood Pressure, in both no apneic and apneic oxygenation application cases are expected.
Comparison of changes in Diastolic Blood Pressure, between first and second tracheal dilatation procedure in children | Changes in Diastolic Blood Pressure between end and start of first/second tracheal balloon dilatation procedure in children
  Evaluation of changes in Diastolic Blood Pressure between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 2nd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Diastolic Blood Pressure between 1st and 2nd tracheal balloon dilatation in children. No significant changes in Systolic Blood Pressure, in both no apneic and apneic oxygenation application cases are expected.
Comparison of changes in Diastolic Blood Pressure, between first and third tracheal dilatation procedure in children | Changes in Diastolic Blood Pressure between end and start of first/third tracheal balloon dilatation procedure in children
  Evaluation of changes in Diastolic Blood Pressure between end and start of 1st tracheal dilatation procedure in children, where no external apneic oxygen enrichment is applied, between end and start of 3rd dilatation procedure, where apneic oxygenation is applied, and comparison of changes in Diastolic Blood Pressure between 1st and 3rd tracheal balloon dilatation in children. No significant changes in Systolic Blood Pressure, in both no apneic and apneic oxygenation application cases are expected.

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Iordanidou, Consultant, Principal Investigator — Hippokratio General Hospital, Thessaloniki, Greece
Locations (1):
- Hippokratio General Hospital, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Overmann KM, Boyd SD, Zhang Y, Kerrey BT. Apneic oxygenation to prevent oxyhemoglobin desaturation during rapid sequence intubation in a pediatric emergency department. Am J Emerg Med. 2019 Aug;37(8):1416-1421. doi: 10.1016/j.ajem.2018.10.030. Epub 2018 Oct 18. PMID 30401594
- [Background] Soneru CN, Hurt HF, Petersen TR, Davis DD, Braude DA, Falcon RJ. Apneic nasal oxygenation and safe apnea time during pediatric intubations by learners. Paediatr Anaesth. 2019 Jun;29(6):628-634. doi: 10.1111/pan.13645. Epub 2019 Apr 29. PMID 30943324
- [Result] Brown SB, Hedlund GL, Glasier CM, Williams KD, Greenwood LH, Gilliland JD. Tracheobronchial stenosis in infants: successful balloon dilation therapy. Radiology. 1987 Aug;164(2):475-8. doi: 10.1148/radiology.164.2.3602388.
- [Result] Cohen MD, Weber TR, Rao CC. Balloon dilatation of tracheal and bronchial stenosis. AJR Am J Roentgenol. 1984 Mar;142(3):477-8. doi: 10.2214/ajr.142.3.477. No abstract available. PMID 6607627
- [Result] Maresh A, Preciado DA, O'Connell AP, Zalzal GH. A comparative analysis of open surgery vs endoscopic balloon dilation for pediatric subglottic stenosis. JAMA Otolaryngol Head Neck Surg. 2014 Oct;140(10):901-5. doi: 10.1001/jamaoto.2014.1742. PMID 25170960
- [Result] Whigham AS, Howell R, Choi S, Pena M, Zalzal G, Preciado D. Outcomes of balloon dilation in pediatric subglottic stenosis. Ann Otol Rhinol Laryngol. 2012 Jul;121(7):442-8. doi: 10.1177/000348941212100704. PMID 22844863
- [Result] Hautefort C, Teissier N, Viala P, Van Den Abbeele T. Balloon dilation laryngoplasty for subglottic stenosis in children: eight years' experience. Arch Otolaryngol Head Neck Surg. 2012 Mar;138(3):235-40. doi: 10.1001/archoto.2011.1439. Epub 2012 Feb 20. PMID 22351854
- [Result] Lang M, Brietzke SE. A systematic review and meta-analysis of endoscopic balloon dilation of pediatric subglottic stenosis. Otolaryngol Head Neck Surg. 2014 Feb;150(2):174-9. doi: 10.1177/0194599813510867. Epub 2013 Nov 5. PMID 24192289
- [Result] HOLMDAHL MH. Pulmonary uptake of oxygen, acid-base metabolism, and circulation during prolonged apnoea. Acta Chir Scand Suppl. 1956;212:1-128. No abstract available. PMID 13326155
- [Result] Mosier JM, Hypes CD, Sakles JC. Understanding preoxygenation and apneic oxygenation during intubation in the critically ill. Intensive Care Med. 2017 Feb;43(2):226-228. doi: 10.1007/s00134-016-4426-0. Epub 2016 Jun 24. No abstract available. PMID 27342820
- [Result] Ricard JD. Hazards of intubation in the ICU: role of nasal high flow oxygen therapy for preoxygenation and apneic oxygenation to prevent desaturation. Minerva Anestesiol. 2016 Oct;82(10):1098-1106. Epub 2016 May 6. PMID 27152499
- [Result] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Result] Kernisan G, Adler E, Gibbons P, Runions B (1987). Apneic oxygenation in pediatric patients. Anesthesiology; 67(3A).
- [Result] Vukovic AA, Hanson HR, Murphy SL, Mercurio D, Sheedy CA, Arnold DH. Apneic oxygenation reduces hypoxemia during endotracheal intubation in the pediatric emergency department. Am J Emerg Med. 2019 Jan;37(1):27-32. doi: 10.1016/j.ajem.2018.04.039. Epub 2018 Apr 18. PMID 29699900
- [Result] Kolettas A, Grosomanidis V, Kolettas V, Zarogoulidis P, Tsakiridis K, Katsikogiannis N, Tsiouda T, Kiougioumtzi I, Machairiotis N, Drylis G, Kesisis G, Beleveslis T, Zarogoulidis K. Influence of apnoeic oxygenation in respiratory and circulatory system under general anaesthesia. J Thorac Dis. 2014 Mar;6 Suppl 1(Suppl 1):S116-45. doi: 10.3978/j.issn.2072-1439.2014.01.17. PMID 24672687
- [Result] Pek JH, Tan HC, Shen G, Ong YG. Apneic Oxygenation for Emergency Intubations in the Pediatric Emergency Department-A Quality Improvement Initiative. Pediatr Qual Saf. 2020 Feb 13;5(2):e255. doi: 10.1097/pq9.0000000000000255. eCollection 2020 Mar-Apr. PMID 32426623
- [Result] Mortimer T, Burzynski J, Kesselman M, Vallance J, Hansen G. Apneic Oxygenation during Rapid Sequence Intubation in Critically Ill Children. J Pediatr Intensive Care. 2016 Mar;5(1):28-31. doi: 10.1055/s-0035-1568149. Epub 2015 Nov 18. PMID 31110879
- [Result] Scott A, Chua O, Mitchell W, Vlok R, Melhuish T, White L. Apneic Oxygenation for Pediatric Endotracheal Intubation: A Narrative Review. J Pediatr Intensive Care. 2019 Sep;8(3):117-121. doi: 10.1055/s-0039-1678552. Epub 2019 Feb 13. PMID 31404416
- [Result] Kurth CD, Thayer WS. A multiwavelength frequency-domain near-infrared cerebral oximeter. Phys Med Biol. 1999 Mar;44(3):727-40. doi: 10.1088/0031-9155/44/3/015. PMID 10211806
- [Result] Kurth CD, Steven JL, Montenegro LM, Watzman HM, Gaynor JW, Spray TL, Nicolson SC. Cerebral oxygen saturation before congenital heart surgery. Ann Thorac Surg. 2001 Jul;72(1):187-92. doi: 10.1016/s0003-4975(01)02632-7. PMID 11465176
- [Result] Kurth CD, Levy WJ, McCann J. Near-infrared spectroscopy cerebral oxygen saturation thresholds for hypoxia-ischemia in piglets. J Cereb Blood Flow Metab. 2002 Mar;22(3):335-41. doi: 10.1097/00004647-200203000-00011. PMID 11891439
- [Result] Tsuji M, Saul JP, du Plessis A, Eichenwald E, Sobh J, Crocker R, Volpe JJ. Cerebral intravascular oxygenation correlates with mean arterial pressure in critically ill premature infants. Pediatrics. 2000 Oct;106(4):625-32. doi: 10.1542/peds.106.4.625. PMID 11015501